CLINICAL TRIAL: NCT05800574
Title: A Phase II Investigation of Lymphoscintigraphy Directed Elective Neck Radiation for p16+ Favorable Risk Oropharynx Cancer Patients Managed With Primary (Chemo) Radiation
Brief Title: Lymphoscintigraphy Directed Elective Neck Radiation for p16+ Favorable Risk Oropharynx Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Cardinal Health (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-1031; HN-107 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Oropharynx Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (>N1 or single node > 3cm ) (Experimental): More extensive neck involvement or proximity to the midline can qualify a patient in cohort A. Cohort A will have patients with either more than one lymph node adenopathy or 1 lymph node that is large (>3cm).
  Interventions: Radiation: Radiation therapy (5 days for 7 weeks); Drug: Cisplatin
- Cohort B (N0 or N1 <3cm) (Experimental): For Cohort B patients need to have either no lymph nodes or only one lymph node adenopathy, provided it is smaller than 3cm.
  Interventions: Radiation: Radiation therapy (5 days for 6 weeks)

INTERVENTIONS:
Radiation: Radiation therapy (5 days for 7 weeks) — Mon-Fri (5 days for 7 weeks), total 35 fractions over 35 treatment days of radiation therapy (RT)
  Arms: Cohort A (>N1 or single node > 3cm )
Radiation: Radiation therapy (5 days for 6 weeks) — Mon-Fri (5 days for 6 weeks), total 35 fractions over 30 treatment days of RT (two doses 6 hours apart except for the last 6th Friday of the 6 weeks )
  Arms: Cohort B (N0 or N1 <3cm)
Drug: Cisplatin — Cisplatin, 40mg/m2 (weekly for 7 weeks)
  Arms: Cohort A (>N1 or single node > 3cm )

SUMMARY:
This is a prospective, phase II, stratified single arm investigation for favorable prognosis in p16+ oropharynx cancer patients with either node negative or malignant neck adenopathy with lymphoscintigraphy mapping confined to the ipsilateral neck.

DETAILED DESCRIPTION:
This is a prospective, phase II, stratified single arm investigation for favorable prognosis in p16+ oropharynx cancer patients with either node negative or malignant neck adenopathy with lymphoscintigraphy mapping confined to the ipsilateral neck. Patients positive for p16 status will be approached for consent during the pre-treatment intake process. Contralateral neck progression will be measured by PET (positron emission tomography)/CT scans. Xerostomia will be measured by the EORTC QLQ (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire) H&N35 at 6, 12, and 24 months. Patients will remain on study treatment for 6-7 weeks or until unacceptable toxicity or withdrawal of consent. Disease free survival (DFS) and overall survival (OS) will be assessed until 24 months after completion of study treatment

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed squamous cell carcinoma of the oropharynx
* Patients to be treated with bilateral neck radiation per current guidelines must have either present (see below):
* Nodal status (based on staging manual, AJCC (American Joint Committee on Cancer) 8th ed.): N0 (provided the tumor is within 1cm of midline) N1> 1 lymph nodes (on the same side of the neck as the primary cancer) or cN3 (cranial nerve III) with no contralateral neck adenopathy
* Tumor stage T1-2 that approaches within 1 cm but does not cross midline as appreciated radiographically and/or by the treating radiation oncologist or a head and neck surgeon
* CT with contrast and/or MRI with contrast performed within 56 days prior to registration that does not demonstrate bilateral neck adenopathy. In the setting of medical contraindication to both CT and MRI contrast please contact the study PI
* PET/CT performed with 28 days prior to registration that does not demonstrate bilateral neck adenopathy.
* Immunohistochemical staining for p16 that demonstrates moderate to severe staining in at least 70% of cells.
* Patients must provide their smoking history prior to registration. Number of pack-years = [Frequency of smoking (number of cigarettes per day) x duration of cigarette smoking (years)]/20
* Patients must have clinically and/or radiographically evident disease that can be accurately measured in accordance with RECIST criteria v. 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1 within 56 days prior to registration
* Age ≥ 18 years.
* Adequate hematologic function within 14 days prior to registration
* Adequate renal function within 14 days prior to registration
* Adequate hepatic function within 14 days prior to registration

Exclusion Criteria:

* Tumors that cross midline, regardless of T stage
* N2 adenopathy (bilateral neck adenopathy)
* Gross total excision of the primary site in a diagnostic procedure prior to either imaging and/or physical examination by registering physician.
* p16-negative squamous cell carcinoma
* Definitive clinical or radiologic evidence of metastatic disease or adenopathy below the clavicles
* Prior systemic therapy for the study cancer
* Prior head and neck cancer surgery that involved the neck (includes excisional biopsy)
* Prior radiation therapy to the head and neck that would result in overlap of treated fields
* History of allergic reaction attributed to Technetium-99m-tilmanocept used in lymphoscintigraphy
* Uncontrolled intercurrent illness including, but not limited to, any other malignancy, other ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-09-23 (Estimated); Study Completion 2027-09-23 (Estimated)

PRIMARY OUTCOMES:
Number of patients that develop cancer on the contra-lateral side of the neck within 12 months of completion of radiation treatment | 1 year
  To evaluate the development of cancer on the contra-lateral side of the neck within 12 months of completion of radiation treatment.

SECONDARY OUTCOMES:
Level of xerostomia | 2 years
  To evaluate whether the omission of elective radiation to the contralateral neck decrease patient reported xerostomia at 6, 12, and 24 months to a mean score of 47.2 (from an expected 57.2) as measured by the European Organization for Research and Treatment of Cancer (EORTC) QLQ H&N35
Mean swallowing change (modified barium swallowing test) | 2 years
  To evaluate the functional swallowing change of patients treated with unilateral neck radiation as measured by a modified barium swallow for the period of one year after the end of radiotherapy. The investigators will use summary statistics such as changes in means and changes in proportions to evaluate the functional swallowing change of patients treated with unilateral neck radiation as measured by a modified barium swallow test.
Mean swallowing change (patient reported) | 2 years
  To evaluate patient reported swallowing of patients treated with unilateral neck radiation as measured by the EORTC QLQ H&N 35 for the period of two years after the end of radiotherapy. The investigators will use summary statistics to characterize changes in means of reported swallowing for patients treated with unilateral neck radiation as measured by the EORTC QLQ H&N 35. The investigators will use sign-rank tests to investigate if the changes are equal to zero.
Rate of contralateral neck progression | 2 years
  To evaluate the development of cancer on the contra-lateral side of the neck within 24 months of completion of radiation treatment. The investigators will use cumulative incidence curves and Fine and Gray proportional hazards regressions to characterize the rate of contralateral neck progression for the period of 2 years after the completion of radiation. In this analysis, death will be considered a competing risk.
Overall survival (OS) | 2 years
  To evaluate the OS of head and neck cancer patients treated with unilateral neck radiation for the period of two years after the end of radiotherapy using Kaplan Meier curves and Cox proportional hazards regressions.
Disease free survival (DFS) | 2 years
  To evaluate the DFS in accordance with RECIST 1.1 of head and neck cancer patients treated with unilateral neck radiation for the period of two years after the end of radiotherapy using Kaplan Meier curves and Cox proportional hazards regressions.
Dosimetric degree of normal tissue avoidance | 2 years
  To quantify the dosimetric degree of normal tissue avoidance of unilateral neck radiation when compared to bilateral neck radiation using Wilcoxon Rank-Sum tests

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Galloway, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No